CLINICAL TRIAL: NCT04229680
Title: The Salty Gut: Effects of High Dietary Salt Intake on the Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1423170
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Cardiovascular Risk Factor
Keywords: Dietary sodium; Gut microbiota

STUDY DESIGN:
Intervention Model Description: All participants will complete each arm.
Who Masked: Participant
Masking Description: Single-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Salt (Experimental): Subjects will be counseled to consume a diet with 2,300 mg/d sodium which they will supplement with pills containing salt to achieve an intake of 6,900 mg/d sodium.
  Interventions: Other: High Salt
- Recommended Salt (Placebo Comparator): Subjects will be counseled to consume a diet with 2,300 mg/d sodium which they will supplement with placebo pills.
  Interventions: Other: Recommended Salt

INTERVENTIONS:
Other: High Salt — Consumption of pills containing table salt for 10 days.
  Arms: High Salt
Other: Recommended Salt — Consumption of pills containing dextrose for 10 days.
  Other Names: Placebo
  Arms: Recommended Salt

SUMMARY:
Gut microbiota has a role in cardiovascular disease and recent findings in rodents show dietary salt can negatively alter gut microbiota composition. High salt intake is a risk factor for cardiovascular disease. Americans consume dietary salt in excess of Dietary Guidelines and American Heart Association recommendations. The objective of this project is to investigate the influence of high dietary salt consumption on the gut microbiota composition in men and women.

DETAILED DESCRIPTION:
Gut microbiota composition and function has an important role in host physiology. In general, gut microbial diversity is positively correlated with health status. Recent evidence confirms the role of gut dysbiosis in cardiovascular disease. Americans consume 50% more salt than the amount recommended by the Dietary Guidelines and 130% more than recommended by the American Heart Association. Excess salt intake is considered a modifiable risk factor for cardiovascular disease. Changes in the gut microbiota composition followed by immune system activation is reported with high salt intake in animals. In particular, abundance of proinflammatory T helper 17 (Th17) cells increases with excess salt consumption. In contrast, T regulatory (Treg) cells oppose Th17 cell action and may aid in reducing inflammation associated with high salt intake, a hypothesis that has not yet been tested in humans. Only one preliminary study assessed changes in gut bacterial composition with high salt intake in humans, when only men were recruited. The study also found an increase in Th17 cell abundance. Thus, the objective of this study is to investigate the influence of high salt intake on the gut microbiota diversity and Th17 and Treg cell abundance in men and women.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* normal blood pressure

Exclusion Criteria:

* hypertension
* cardiovascular disease
* renal disease
* diabetes
* cancer
* current use of anti-inflammatory agents, glucocorticoids or other immune regulating medications, or certain anti-depressants
* history of intestinal surgery
* inflammatory bowel disease, celiac disease, lactose intolerance, chronic pancreatitis or other malabsorption disorder
* antibiotic use in the past 3 months
* prebiotic, probiotic, or antioxidant supplementation in the past 3 months
* ≥10 lbs weight gain or loss in the past 6 months
* use of tobacco products
* highly trained endurance athletes
* current pregnancy or lactation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Gut microbiota diversity | On day 10
  The difference in gut microbiota diversity between the two arms.
T cell profile | On day 10
  The difference in T regulatory and T helper 17 cells between each arm.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon L Lennon, PhD, RD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States